CLINICAL TRIAL: NCT06937814
Title: The Effect of Humiome® Post LB on Gut COMFort in healthY Adult Volunteers: a Double-blind, Randomized Placebo-controlled Study
Brief Title: The Effect of Humiome® Post LB on Gut COMFort in healthY Adult Volunteers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-10-24-POSTL
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: GI Issues; Bowel Movements; Gastrointestinal Symptoms
Keywords: Bowel movements; Gastrointestinal symptoms; Bristol stool scale

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Humiome® Post LB (Experimental): A postbiotic comprised of inactivated Limosilactobacillus fermentum (CNCM I-2998) and Lactobacillus delbrueckii (CNCM I-4831), together referred to as Lactobacillus LB, and fermented culture medium.
  Interventions: Dietary Supplement: Humiome ® Post LB
- Placebo (Placebo Comparator): 170 mg/day of micro-crystalline cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Humiome ® Post LB — Participants will be instructed to take one capsule with a glass of water after the first meal of the day.
  Arms: Humiome® Post LB
Other: Placebo — Participants will be instructed to take one capsule with a glass of water after the first meal of the day.
  Arms: Placebo

SUMMARY:
The goal of this double-blind, randomized placebo-controlled study is to evaluate the effect of an 8-week supplementation of Humiome ® Post LB (170 mg) on bowel movements in healthy adult volunteers compared to Placebo adjusted on baseline. The main question[s] it aims to answer [is/are]:

Does Humiome ® Post LB improve bowel movements with self-reported GI issues?

Participants will be provided Humiome ® Post LB (170 mg) for 8 weeks and asked to complete a study diary, questionnaires, and stool samples.

ELIGIBILITY:
Inclusion Criteria:

1. Be able to give written informed consent.
2. Self-reported gastrointestinal issues defined as 10-20 bowel movements per week and a score of 5-6 for ≥20% of stools based on the BSS in the 2 weeks prior to baseline, as assessed by the Qualified Investigator (QI).
3. Self-reported GI issues such as bloating, mild cramping, and urgency, as assessed by the QI.
4. Be between 18 and 75 years of age, inclusive.
5. Have a BMI of between 18.5 - 29.9 kg/m2, inclusive.
6. Self-reported stable body weight (<5% change) over the past 3 months.
7. Be in general good health, as determined by the QI.
8. Willing to avoid consuming prebiotic, probiotic, postbiotics, fiber-rich and dietary supplements, anti-diarrheal and anti-constipation medication until the end of the study (see Section 5.6).
9. Willing to maintain current dietary habits and lifestyle, including level of physical activity, allowed medication/supplements habits for the duration of the study.
10. Females not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening Or,

Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method
* Intrauterine devices
* Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
* Vasectomy of partner at least 6 months prior to screening
* Abstinence and agrees to use contraception if planning on becoming sexually active during the study

Exclusion Criteria:

1. Failure to meet any one of the inclusion criteria.
2. Females who are pregnant, lactating or wish to become pregnant during the study.
3. Are lactose intolerant or have any other hypersensitivity/allergy to any of the components of the test product.
4. Meeting Irritable Bowel Syndrome (IBS) diagnostic criteria as defined by Rome IV criteria, i.e. having recurrent abdominal pain on average at least 1 day/week in the last 3 months, associated with two or more of the following criteria:

   1. Related to defecation.
   2. Associated with a change in frequency of stool.
   3. Associated with a change in form (appearance) of stool. Criteria need to be fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis.
5. Have suffered from diarrhea (defined as ≥3 bowel movements per day and 6-7 on BSS) at any time two weeks prior to run-in, as assessed by the QI.
6. Experience alarm features such as weight loss, rectal bleeding, or recent change in bowel habit (<3 months), as assessed by the QI.
7. Have taken antibiotics within the previous 2 months prior to the run-in period as assessed by QI (see Section 5.6.1).
8. Unstable hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg). Treatment on a stable dose of medication for at least 3 months will be considered by the QI.
9. Known history of or ongoing HIV, hepatitis or clinically important, as judged by the QI, endocrine (including Type 1 or Type 2 diabetes mellitus), cardiovascular (including, but not limited to, atherosclerotic disease, history of myocardial infarction, peripheral arterial disease, stroke), pulmonary, biliary conditions.
10. Current or history of any significant diseases of the gastrointestinal tract (including but not limited to Crohn's disease, ulcerative colitis, celiacs disease, colectomy), as assessed by the QI.
11. Have planned a major surgery during the study period as assessed by the QI.
12. Have a history of drug and/or alcohol abuse in the past 12 months at the time of enrolment.
13. Alcohol intake average of >2 standard drinks per day as assessed by the QI
14. Have made any major dietary changes in the past 3 months prior to run-in period.
15. Currently consuming a vegetarian or vegan diet.
16. Are planning a holiday over the study period that would alter dietary patterns as assessed by the QI.
17. Have planned major changes in lifestyle (i.e. diet, weight loss program, exercise level, travelling) during the duration of the study.
18. Regular use of tobacco or nicotine products in the past six months, as assessed by the QI. Occasional users will be required to washout and abstain for the duration of the study period.
19. Chronic use of cannabinoid products (>2 times/week). Occasional users will be required to abstain for the duration of the study period.
20. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant.
21. Participation in other clinical research studies 30 days prior to the run-in period, as assessed by the QI.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of Humiome ® Post LB (170 mg) supplementation on bowel movements in healthy adult volunteers compared to Placebo | Day 0 to 56
  To evaluate the effect of Humiome ® Post LB (170 mg) supplementation on the difference in frequency of bowel movements as assessed by the Bowel Habits Diary (BHD) in healthy adult volunteers compared to Placebo adjusted on baseline at week 8 (Day 56; between group comparison).

SECONDARY OUTCOMES:
The difference in frequency of bowel movements between Humiome® Post LB and Placebo | Day 0 to 28
  The difference in frequency of bowel movements as assessed by the BHD at week 4 (Day 28) between Humiome® Post LB and Placebo
The difference in frequency of bowel movements after Humiome® Post LB and Placebo compared to baseline. | Day 0 to 28
  The difference in frequency of bowel movements as assessed by the BHD after Humiome® Post LB and Placebo at weeks 4 (Day 28) compared to baseline.
The difference in frequency of bowel movements after Humiome® Post LB and Placebo compared to baseline. | Day 0 to 56
  The difference in frequency of bowel movements as assessed by the BHD after Humiome® Post LB and Placebo at week 8 (Day 56) compared to baseline.
The difference between Humiome® Post LB and Placebo in stool consistency. | Day 0 to 28
  The difference at weeks 4 (Day 28) between Humiome® Post LB and Placebo in stool consistency as assessed by the Bristol Stool Scale.
The difference between Humiome® Post LB and Placebo in stool consistency. | Day 0 to 56
  The difference at weeks 8 (Day 56) between Humiome® Post LB and Placebo in stool consistency as assessed by the Bristol Stool Scale
The difference between Humiome® Post LB and Placebo in quality of life | Day 0 to 28
  The difference at weeks 4 (Day 28) between Humiome® Post LB and Placebo in quality of life as assessed by the RAND Short Form Health Survey 36 (SF-36).
The difference between Humiome® Post LB and Placebo in quality of life | Day 0 to 56
  The difference at weeks 8 (Day 56) between Humiome® Post LB and Placebo in quality of life as assessed by the RAND Short Form Health Survey 36 (SF-36).
The difference after Humiome® Post LB and Placebo compared to baseline in stool consistency | Day 0 to 28
  The difference after Humiome® Post LB and Placebo at weeks 4 (Day 28) compared to baseline in stool consistency as assessed by the Bristol Stool Scale
The difference after Humiome® Post LB and Placebo compared to baseline in stool consistency | Day 0 to 56
  The difference after Humiome® Post LB and Placebo at weeks 8 (Day 56) compared to baseline in stool consistency as assessed by the Bristol Stool Scale
The difference after Humiome® Post LB and Placebo compared to baseline in quality of life | Day 0 to 28
  The difference after Humiome® Post LB and Placebo at weeks 4 (Day 28) compared to baseline in quality of life as assessed by the RAND Short Form Health Survey 36 (SF-36).
The difference after Humiome® Post LB and Placebo compared to baseline in quality of life | Day 0 to 56
  The difference after Humiome® Post LB and Placebo at weeks 8 (Day 56) compared to baseline in quality of life as assessed by the RAND Short Form Health Survey 36 (SF-36).
The difference between Humiome® Post LB and Placebo in fecal microbial composition | Day 0 to 56
  The difference at week 8 (Day 56) between Humiome® Post LB and Placebo in fecal microbial composition (i.e., relative abundance of taxa) as assessed by shallow shotgun sequencing.
The difference between Humiome® Post LB and Placebo in fecal microbial composition | Day 0 to 56
  The difference at week 8 (Day 56) between Humiome® Post LB and Placebo in fecal bacterial diversity as assessed by shallow shotgun sequencing.
The difference after Humiome® Post LB and Placebo compared to baseline in fecal microbial composition | Day 0 to 56
  The difference after Humiome® Post LB and Placebo at week 8 (Day 56) compared to baseline in fecal microbial composition (i.e., relative abundance of taxa) as assessed by shallow shotgun sequencing.
The difference after Humiome® Post LB and Placebo compared to baseline in fecal bacterial diversity | Day 0 to 56
  The difference after Humiome® Post LB and Placebo at week 8 (Day 56) compared to baseline in fecal bacterial diversity as assessed by shallow shotgun sequencing.

OTHER OUTCOMES:
The difference between Humiome® Post LB and Placebo in GI symptoms | Day 0 to 28
  The difference at weeks 4 (Day 28) between Humiome® Post LB and Placebo in GI symptoms as assessed by the Gastrointestinal Symptom Rating Scale (GSRS)
The difference between Humiome® Post LB and Placebo in GI symptoms | Day 0 to 56
  The difference at weeks 8 (Day 56) between Humiome® Post LB and Placebo in GI symptoms as assessed by the Gastrointestinal Symptom Rating Scale (GSRS)
The difference after Humiome® Post LB and Placebo compared to baseline in GI symptoms | Day 0 to 28
  The difference after Humiome® Post LB and Placebo at weeks 4 (Day 28) compared to baseline in GI symptoms as assessed by the Gastrointestinal Symptom Rating Scale (GSRS)
The difference after Humiome® Post LB and Placebo compared to baseline in GI symptoms | Day 0 to 56
  The difference after Humiome® Post LB and Placebo at weeks 8 (Day 56) compared to baseline in GI symptoms as assessed by the Gastrointestinal Symptom Rating Scale (GSRS)
The difference after Humiome® Post LB and Placebo in perceived benefits | Day 0 to 56
  The difference at week 8 (Day 56) between Humiome® Post LB and Placebo in perceived benefits as assessed by a 5-point Likert scale
To evaluate in healthy volunteers the effect of daily consumption of 170 mg Humiome® Post LB on safety variables | Day 0 to 56
  To evaluate in healthy volunteers the effect of daily consumption of 170 mg Humiome® Post LB on adverse events and serious adverse events.
Clinically relevant changes in blood pressure | Day 0 to 56
  Clinically relevant changes in blood pressure (BP) after supplementation from baseline (visit 2) at end of the study (visit 4).
Clinically relevant changes in heart rate | Day 0 to 56
  Clinically relevant changes in heart rate after supplementation from baseline (visit 2) at end of the study (visit 4).

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No